CLINICAL TRIAL: NCT03672019
Title: Health-Related Quality of Life in Patients Undergoing Percutaneous Biliary Drainage For Malignant Biliary Obstruction
Brief Title: A Quality of Life Study in Patients Undergoing Percutaneous Biliary Drainage
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 18-366
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Malignant Biliary Obstruction
Keywords: Percutaneous Biliary Drainage; Quality of life; 18-366

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Undergoing Percutaneous Biliary Drainage: Following Percutaneous Biliary Drainage (PBD), participants will complete Patient Reported Outcomes (PRO) assessments at baseline and at three time points post-procedure: 4 weeks (+/- 1 weeks), 12 weeks (+/- 2 weeks), and 6 months (+/- 2 weeks).
  Interventions: Behavioral: FACT-Hep

INTERVENTIONS:
Behavioral: FACT-Hep — Patient Reported Outcomes (PRO) assessments at baseline and at three time points post-procedure: 4 weeks (+/- 1 weeks), 12 weeks (+/- 2 weeks), and 6 months (+/- 2 weeks).
  Other Names: The Functional Assessment of Cancer Therapy

SUMMARY:
The purpose of this study is to compare the participant's health-related quality of life before and after the biliary drainage procedure. The study will also help us learn whether having a drainage catheter or a stent placed during the procedure makes a difference in the participant's quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known malignancy presenting for treatment of biliary obstruction
* Undergoing initial Interventional Radiology PBD procedure
* Fluent in English to enable instrument completion
* At least18 years of age
* Must be physically and mentally capable of completing instruments
* Must be able to comprehend and execute informed consent

Exclusion Criteria:

* Patients will be excluded if:

  * Indication for drainage is acute, symptomatic cholangitis requiring an emergent procedure
  * Previous PBD procedure
  * Presence of an indwelling biliary stent
* Medical or psychiatric condition that, in the judgment of the consenting professional, prevents appropriate comprehension and execution of either the informed consent or the study instruments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified in the interventional radiology clinic or while admitted based on a request for a biliary drainage procedure from their primary oncologist or surgeon at MSK.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
change in the FACT-Hep scores | baseline to week 4 post-procedure
  The FACT-Hep minimum score is 0 and the maximum is 180.

CONTACTS AND LOCATIONS:
Overall Officials: Piera Cote Robson, MSN, CNS, NP, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm